CLINICAL TRIAL: NCT02732782
Title: Effectiveness of Eccentric Exercise Compared to Isometric Exercise in Athletes With Chronic Achilles Tendinopathy
Brief Title: Effectiveness of Isometric vs. Eccentric Exercise in Chronic Achilles Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Humboldt-Universität zu Berlin (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Goran Radovanovic, Principal Investigator, Humboldt-Universität zu Berlin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR020151100167; AZ: ZMV14-070102/16-17 (Other Grant/Funding Number: Bundesinstitut für Sportwissenschaft (BISp))
Record Dates: First submitted 2016-03-22; First posted 2016-04-11 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Tendinopathy
Keywords: Achilles tendon; isometric muscle training; competitive sports; strength training; eccentric exercise; isometric exercise; chronic condition; regeneration; tendon; tendon properties; tendinopathy; tendinosis; intervention; training load; high performance sports
MeSH Terms: conditions — Tendinopathy; Chronic Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Isometric exercise (Experimental): Isometric exercise (90% maximum voluntary contraction (MVC), 12 weeks, 4 times a week, 5 sets of 4 repetitions a 3 seconds)
  Interventions: Other: Isometric exercise
- Eccentric exercise (Active Comparator): Eccentric training ("Alfredson" approach, 12 weeks, 2 sets per day with extended and two sets per day with bended knee, 15 repetitions per set)
  Interventions: Other: Eccentric exercise
- Control (No Intervention): Control, no intervention

INTERVENTIONS:
Other: Isometric exercise
  Arms: Isometric exercise
Other: Eccentric exercise
  Arms: Eccentric exercise

SUMMARY:
This is a prospective single blinded randomised controlled trial with a 12-week intervention period and a half-year follow-up period. The main purpose is to determine the effects of isometric exercise on mechanical, morphological and functional tendon properties versus eccentric exercise in chronic Achilles tendinopathy.

DETAILED DESCRIPTION:
This research project was funded by means of the "Bundesinstitut für Sportwissenschaft" based on a resolution of the German Federal Parliament.

ELIGIBILITY:
Inclusion Criteria:

* Chronic (3 months or more) condition of unilateral Achilles tendinopathy confirmed by a medical doctor based on ultrasound
* age 18-60
* male
* VISA-A Score of at least 80

Exclusion Criteria:

* bilateral tendinopathy
* any systemic or inflammatory diseases (i. e. Diabetes, Arthritis)
* surgery on lower extremities in the past
* corticoid injections in the last 12 months

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2016-08; Primary Completion 2019-02-28 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Morphological tendon properties, Tendon cross sectional area (CSA) | At baseline and 12 weeks after
  Equipment Magnetic resonance imaging (MRI) (0.25 T MR Scanner (Esaote, G-Scan, Italy), T1-Gewichtung, 3D HYCE (GR) Sequency, TR 10 ms, TE 5 ms, flip angle 80°, layer thickness 3 mm, 1 Anregung) Software OsiriX (Pixmeo SARL, Version 2.5.1., Schweiz)
  Tendon thickness / cross sectional area (CSA) in square millimeter (mm²) through MRI, manually outlined via Software OsiriX (Pixmeo SARL, Version 2.5.1., Schweiz). The mean value of three measurements of the same image will be used for analysis. In order to demonstrate local changes within the tendon, CSA will be shown in 10% intervals relative to the total length of the tendon.
Mechanical tendon properties, Tendon stiffness | At baseline and 12 weeks after
  Equipment Dynamometer (Biodex System 3, Medical Systems Inc., USA), optical motion capture system with eight cameras with a frequency of 250 Hertz (Hz) (Vicon Nexus, version 1.7.1., Vicon Motion Systems, UK), electromyography (Myon m320RX, Myon AG, Schweiz) and a linear ultrasound (7.5 Megahertz (MHz), ESAOTE MyLab 60)
  Tendon stiffness in Newton per mm (N/mm) with support of tendon force in Newton (N)
Mechanical tendon properties, Modulus | At baseline and 12 weeks after
  Equipment Dynamometer (Biodex System 3, Medical Systems Inc., USA), optical motion capture system with eight cameras with a frequency of 250 Hertz (Hz) (Vicon Nexus, version 1.7.1., Vicon Motion Systems, UK), electromyography (Myon m320RX, Myon AG, Schweiz) and a linear ultrasound (7.5 Megahertz (MHz), ESAOTE MyLab 60)
  Modulus in Pascal (Pa) based on tendon stress (Pa) and tendon elongation in millimeter (mm)
Morphological tendon properties, Tendon length | At baseline and 12 weeks after
  Equipment Magnetic resonance imaging (MRI) (0.25 T MR Scanner (Esaote, G-Scan, Italy), T1-Gewichtung, 3D HYCE (GR) Sequency, TR 10 ms, TE 5 ms, flip angle 80°, layer thickness 3 mm, 1 Anregung) Software OsiriX (Pixmeo SARL, Version 2.5.1., Schweiz)
  Tendon length im millimeter (mm) through MRI, manually outlined via Software OsiriX (Pixmeo SARL, Version 2.5.1., Schweiz).The mean value of three measurements of the same image will be used for analysis.
Morphological tendon properties, Tendon vascularization level | At baseline and 12 weeks after
  Equipment Linear ultrasound (7.5 Megahertz (MHz), ESAOTE MyLab 60) Software Doppler Flow Image Analyser version 1.01
  Vascularization level of the tendon via Color Doppler (CD) ultrasound CD signals will be estimated through the total number of coloured pixels within the area of interest (3x7 centimeters (cm) with the help of Software Doppler Flow Image Analyser version 1.01 (http://www.gtech.dk).

SECONDARY OUTCOMES:
Clinical functional score | At baseline, 12 weeks and six months after
  Victorian Institute of Sport (VISA) - Achilles (A) questionnaire scores from 0 points to 100 points.
Interleukin 6 level | At baseline and 12 weeks after
  Interleukin 6 (IL- 6) detection in the blood plasma is measured in picogram per milliliter (pg/ml) unit.
Functional tendon properties, Ground contact time | At baseline and 12 weeks after
  Drop jumps and counter movement jumps on a three dimensional force plate (AMTI, BP400600-2000, 60x40 cm, 1000 Hz)
  Ground contact time is estimated through ground reaction forces (N or kN).
Functional tendon properties, Maximum jump height | At baseline and 12 weeks after
  Drop jumps and counter movement jumps on a three dimensional force plate (AMTI, BP400600-2000, 60x40 cm, 1000 Hz)
  Maximum jump height is estimated through the vertical impulse / component of the ground reaction force in Newton (N) or Kilo Newton (kN)
Pain level via Visual Analogue Scale (VAS) | At baseline, 12 weeks and six months after
  A Visual Analogue Scale (VAS) for pain reaching from 0mm to 100mm as part of the VISA - A questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Legerlotz, PhD, Prof, Study Director — Humboldt Universität zu Berlin, Department of Movement Sciences
Locations (1):
- Humboldt Universität zu Berlin, Institut für Bewegungswissenschaften, Department Movement Sciences, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Legerlotz K, Jones ER, Screen HR, Riley GP. Increased expression of IL-6 family members in tendon pathology. Rheumatology (Oxford). 2012 Jul;51(7):1161-5. doi: 10.1093/rheumatology/kes002. Epub 2012 Feb 15. PMID 22337942
- [Background] Mersmann F, Bohm S, Schroll A, Boeth H, Duda GN, Arampatzis A. Muscle and tendon adaptation in adolescent athletes: A longitudinal study. Scand J Med Sci Sports. 2017 Jan;27(1):75-82. doi: 10.1111/sms.12631. Epub 2015 Dec 8. PMID 26644277
- [Background] Arampatzis A, Karamanidis K, Mademli L, Albracht K. Plasticity of the human tendon to short- and long-term mechanical loading. Exerc Sport Sci Rev. 2009 Apr;37(2):66-72. doi: 10.1097/JES.0b013e31819c2e1d. PMID 19305197
- [Derived] Radovanovic G, Bohm S, Peper KK, Arampatzis A, Legerlotz K. Evidence-Based High-Loading Tendon Exercise for 12 Weeks Leads to Increased Tendon Stiffness and Cross-Sectional Area in Achilles Tendinopathy: A Controlled Clinical Trial. Sports Med Open. 2022 Dec 20;8(1):149. doi: 10.1186/s40798-022-00545-5. PMID 36538166